CLINICAL TRIAL: NCT02173730
Title: Pharmacokinetics of BIBR 953 ZW After 150 mg of BIBR 1048 (Oral Pro-drug of BIBR 953) Administered as Capsule Twice Daily Over Seven Days With or Without Pantoprazole Co-treatment to Healthy Male and Female Elderly Subjects
Brief Title: BIBR 953 ZW in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.10
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Pantoprazole

ARMS (2):
- BIBR 1048 MS without Pantoprazole (Experimental): 150 mg BIBR 1048 MS capsules administered twice daily over 6 days and once in the morning of the seventh day
  Interventions: Drug: BIBR 1048 MS
- BIBR 1048 MS with Pantoprazole (Experimental): 150 mg BIBR 1048 MS capsules administered twice daily over 6 days and once in the morning of the seventh day together with Pantoprazole. Pantoprazole administration (40 mg bid) started two days before administration og BIBR 1048 and ended in the morning of the seventh day.
  Interventions: Drug: BIBR 1048 MS; Drug: Pantoprazole

INTERVENTIONS:
Drug: BIBR 1048 MS — BIBR 1048 MS capsule 150 mg
Drug: Pantoprazole — Pantoprazole tablet 40 mg
  Arms: BIBR 1048 MS with Pantoprazole

SUMMARY:
To assess the steady state pharmacokinetic profile of BIBR 953 ZW after administration of BIBR 1048 to male and female elderly subjects, to assess pharmacokinetic gender differences. To assess the effect of coadministration of Pantoprazole on the bioavailability of BIBR 953 ZW.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female elderly subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 65, no upper limit
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding at the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of relevant orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * cranio-cerebral trauma
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs that might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol intake (>30 - 40 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 140000/μl (male) or < 156000/μl (female)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-11; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the plasma concentration time curve during a dosing interval at steady state) | Day 4 and 7
Cmax,ss (maximum measured concentration of the analyse in plasma at steady state over a uniform dosing interval τ) | Day 4 and 7
Aeτ,ss (amount of dose excreted in urine over one dosing interval at steady state) | Day 4 and 7
feτ,ss (percent of dose excreted in urine over one dosing interval at steady state) | Day 4 and 7
AUC0-tz,ss (area under the plasma concentration time curve (AUC) from zero time (pre dose) to the time of the last quantifiable concentration (tz)) | Day 4 and 7
Cmin,ss (minimum measured concentration of the analyse in plasma at steady state over a uniform dosing interval τ) | Day 4 and 7
tmax,ss (time from last dosing to the maximum concentration of the analyse in plasma at steady state over a uniform dosing interval τ) | Day 4 and 7
t½,ss (terminal half-life, calculated from the terminal elimination rate constant) | Day 4 and 7

SECONDARY OUTCOMES:
CLR,ss (renal clearance at steady state following multiple dose administration) | Day 4 and 7
MRTss (steady state mean residence time) | Day 4 and 7
CL/F,ss (apparent clearance of the analyse in plasma at steady state after extravascular multiple dose administration) | Day 4 and 7
Vz/F,ss (apparent volume of distribution during the terminal phase at steady state following extravascular administration) | Day 4 and 7
Changes in activated partial thromboplastin time (aPTT) | Day 4 and 7
Changes in ecarin clotting time (ECT) | Day 4 and 7
Occurrence of Adverse Events | up to 10 days